CLINICAL TRIAL: NCT04027504
Title: A Study to Evaluate the Palatability of a Nutritional Support Biscuit (Fitabisc) in Patients About to Undergo Abdominal Surgery
Brief Title: Palatability of Antioxidant Biscuits
Acronym: Fitabisc2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The biscuits contain higher than the UK recommended daily dose of vitamins C and E, and selenium.
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2206
Record Dates: First submitted 2019-06-26; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Preoperative Care; Antioxidants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fitabisc (Experimental): Participants receiving fitabisc preoperatively
  Interventions: Dietary Supplement: Fitabisc

INTERVENTIONS:
Dietary Supplement: Fitabisc — Biscuits containing antioxidants

SUMMARY:
Patients who are due to have planned bowel surgery will be invited to take part in the study. Those that consent, will be given a 5 day supply of 'Fitabisc' (a biscuit designed to have the potential to provide nutritional support).Participants will be asked to eat 4 biscuits a day for a minimum of 5 days prior to their surgery before they are admitted to hospital. They will be asked to complete questionnaires to record the palatability of the biscuit, how much of the daily amount they were able to eat and if they could not eat the full amount, the reason for this.

Information will also be collected on patient's demographic and clinical details.

We will follow participants' progress after surgery so we can be alerted to any possible medium to longer term adverse effects of eating the biscuit, though none are expected.

DETAILED DESCRIPTION:
Nutrition and diet have been shown to have a direct impact on the health of the population and of selected patient groups. These beneficial effects have been attributed to the reduction of oxidative damage caused by the normal or excessive free radical production.

Antioxidants (AOX) are substances which inhibit or delay oxidation. The most important source of AOX is dietary intake. The trace elements copper, selenium, manganese, and zinc are all essential components of endogenous AOX defences. Nutritional antioxidants act through different mechanisms but are mainly free radical scavengers.

Oxidative stress occurs when there is an imbalance between generation of reactive oxygen species and inadequate antioxidant defence systems. Oxidative stress can cause cell damage either directly or through altering signalling pathways. Oxidative stress is a unifying mechanism of injury in many types of disease processes, including gastrointestinal diseases. Not surprisingly, many studies have investigated the potential clinical benefits of administering AOX to various patient groups. These results indicate that AOX nutrients do have a role in the intracellular prevention of AOX related damage and of proximity damage propagation. AOX, in particular appear effective in reducing damage which occurs as a result of ischaemia reperfusion injury.

The evidence suggests that the timing of AOX supplementation is important. It is unlikely that AOX will be able to reverse pathological change but they may limit its extension. In acute conditions the concept of a therapeutic window is essential. There appears to be an optimal early timing during which supplementation may have a "preventative" effect. The magnitude of this is probably determined by premorbid state. It is interesting to speculate, therefore, that pre loading with AOX might mitigate against severity of oxidative damage following a defined injury including surgery. There are theoretical reasons to consider that preoperative antioxidant therapy may be beneficial however there are no data available to date that confirms benefits in clinical practice and in particular as a preoperative supplement. Most studies to date have looked perioperative or postoperative supplementation with the antioxidants alone. No attempt has been made to do this using a palatable biscuit that would facilitate preoperative oral supplementation.

The rationale for this study is to establish whether or not Fitabisc, a biscuit that contains key antioxidants can be tolerated for up to 5 days before surgery in patients undergoing abdominal operations.

If this study confirms palatability and adherence to eating the biscuit then it would be our aim to set up a prospective randomised study in which the potential efficacy of Fitabisc would be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 16 and 90 years
* Having planned abdominal surgery at Castle Hill Hospital

Exclusion Criteria:

* People who do not give informed consent
* People with a known or suspected allergy to gluten and / or dairy products
* People already taking any of the following as dietary supplements: vitamins C, E, selenium or glutamine
* People with haemochromatosis, thalassaemia, kidney disease, liver disease or Reye syndrome
* People with type 1 diabetes or people with type 2 diabetes who take insulin or hypoglycaemic drugs such as Metformin

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-09-20 (Estimated); Study Completion 2018-12-20 (Estimated)

PRIMARY OUTCOMES:
Palatibility Test | 10 days prior to surgery
  Do patients about to undergo colorectal surgery find Fitabisc sufficiently palatable that they can eat the biscuit in the required quantities for 10 days prior to their surgery?

CONTACTS AND LOCATIONS:
Overall Officials: John Hartley, MD FRCS, Principal Investigator — Hull and East Yorkshire NHS Trust
Locations (1):
- Castle Hill Hospital, Hull, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No